CLINICAL TRIAL: NCT00787410
Title: An Open-label, Phase II Trial of ZD1839 (IRESSA) in Patients With Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0094
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Mesothelioma
Keywords: malignant mesothelioma; IRESSA; ZD1839
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ZD1839

INTERVENTIONS:
Drug: ZD1839 — 250mg tablet, once daily, orally administered
  Other Names: IRESSA

SUMMARY:
This study is a multicentre, open label, non-comparative, two stage phase II trial to assess the activity of ZD1839 (IRESSA) in patients with malignant mesothelioma. Patients will receive trial treatment as first-line therapy, administered continuously once daily until the completion of six 4-week cycles of treatment, disease progression, unacceptable toxicity or withdrawal of consent. Patients continuing to show evidence of response, disease stabilization or clinical benefit from ZD1839 may continue to receive therapy beyond completion of the trail.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed malignant mesothelioma (based on pleural biopsy); eligibility for first line therapy for malignant mesothelioma
* Uni or bi- dimensionally measurable disease
* No prior radiotherapy within 3 weeks of enrolment into the trial
* No significant comorbid disease

Exclusion Criteria:

* Other malignancies, either co-existing or diagnosed within the last 5 years, with the exception of basal cell carcinoma or cervical cancer in situ
* Brian metastasis or leptomeningeal carcinomatosis
* Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, or St. John's Wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To assess the activity of ZD1839 in patients with malignant mesothelioma by estimating the objective response rate (CR and PR) at trial closure | Proportion of patients responding at trial closure, ITT population
To further characterize the safety profile of ZD1839 at a 250mg daily dose | Proportion of patients responding at trial closure, ITT population

SECONDARY OUTCOMES:
To estimate PFS (progression free survival) | Proportion of patients alive and progression-free at trial closure, ITT population; Median time to progression or death; Proportion of patients alive and progression-free at 6 months
To estimate overall survival | Proportion of patients alive at trial closure, ITT population; Median time to death; Proportion of patients alive at 6 months
To estimate duration of response | Median time from objective response to progression or death; only patients who responded are included in this analysis

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lee, MD, Principal Investigator — Fraser Valley Cancer Centre Surrey Memorial Hospital, Surrey BC, Canada